CLINICAL TRIAL: NCT05006222
Title: Effects of Enzyme Replacement Therapy on Quality of Life, Functional Independence and Aerobic Capacity in Children With Mucopolysaccharidosis
Brief Title: The Effect of Enzyme Replacement Therapy in Mucopolysaccharidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Assistant of professeur, Hasan Kalyoncu University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020/117
Record Dates: First submitted 2021-08-04; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Mucopolysaccharidosis
Keywords: Mucopolysaccharidosis; Aerobic capacity; Quality of Life; Functional independence
MeSH Terms: conditions — Mucopolysaccharidoses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERT group (Active Comparator): The participants are enrolled in this group whose get enzyme replacement therapy
  Interventions: Drug: Enzyme Replacement Agent
- non-ERT group (No Intervention): The participants are enrolled in this group whose not get enzyme replacement therapy

INTERVENTIONS:
Drug: Enzyme Replacement Agent — Enzyme replacement therapy is one such treatment and used for the management of some subtypes of MPS disease. Enzyme replacement therapy (ERT) is based on the concept of replacing the missing enzyme in the circulation to prevent the build-up of glycosaminoglycan (GAG) in the tissues
  Arms: ERT group

SUMMARY:
Mucopolysaccharidosis (MPS) causes chronic, progressive systemic disorders due to enzyme deficiency. Musculoskeletal manifestations of MPS include bone and vertebral deformities, restricted joint function and ROM (range of motion), rib cage abnormalities, short stature and hip dysplasia as well as flexion contracture in the knee and interphalangeal joints and joint laxity. Currently, there is no treatment that cures the symptoms of MPS. However, there are some forms of treatment that can delay the progression of the disease. Enzyme replacement therapy is one such treatment and used for the management of some subtypes of MPS disease. Enzyme replacement therapy (ERT) is based on the concept of replacing the missing enzyme in the circulation to prevent the build-up of glycosaminoglycan (GAG) in the tissues. Very few studies in the literature have examined the impact of MPS in the lives of children affected by this disease. Studies investigating functional capacity, independence and quality of life in children receiving or not receiving enzyme replacement therapy have not provided a clear picture of the problems faced by these children. Secondly, psychological problems experienced by caregivers of children with MPS have not been studied specifically in former studies. Therefore, the aim of this study was to examine the impact of ERT on aerobic capacity, functional independence and quality of life in children with MPS and to determine the anxiety and depression levels of their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Age must be range between 3 and 11 years
* Having diagnosis of MPS.

Exclusion Criteria:

* Patients refusing to participate in the study
* Patients without a definite diagnosis
* Patients and parents who are not cooperate with the study tests

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-27 (Actual)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory | 1 year
  The Pediatric Quality of Life Inventory (PedsQL) is a health status instrument for the assessment of health-related quality of life in children and adolescents from 2 to 18 years of age. The PedsQL can be completed by children themselves or with their parents. The tool consists of a total of 23 questions that assess physical functioning (8 questions), emotional functioning (5 questions), social functioning (5 questions), and school functioning (5 questions). Possible maximum scores range between 0 and 100 and higher scores indicate better quality of life.
Functional Independence Measure | 1 year
  Functional independence of the subjects was assessed using the Functional Independence Measure for Children (WeeFIM). It is a short and validated tool to determine impairment of developmental, educational and social functioning in children with cerebral palsy and other developmental disorders. The WeeFIM is an 18-item scale that measures the performance of the child in activities of daily living including bowel and bladder control, transfers, mobility, communication, eating, grooming, bathing, upper body dressing, lower body dressing, toileting and social cognition. Each item is assigned a score between 1 and 7 points. Higher total scores indicate greater level of independence.
Aerobic Capacity | 1 year
  Aerobic capacity was assessed using the 6-minute walk test (6MWT) and timed up and go (TUG) test. For the 6MWT test, the subjects were asked to walk but not run for 6 minutes on a 30-meter corridor as fast as possible. Care was taken not to change the pace. At the end of the test, total distance covered was measured.
  The TUG test is a practical test that allows quick assessment of dynamic balance, gait speed and mobility. During the test, the subjects were asked to stand up from a chair without holding on to the arms of the chair, walk 3 meters, turn, return to the chair without touching anything and sit down again. Total time was recorded in seconds.

SECONDARY OUTCOMES:
Balance | 1 year
  The modified functional reach test was developed by Lynch et al. to evaluate dynamic balance of the trunk. It is a reliable and validated test to measure the distance an individual can reach forward without losing balance while sitting in a fixed position. For the test, the subjects were instructed to sit with the arm kept parallel to the wall and shoulder flexed to 90 degrees and measurement was taken from the distal end the third metacarpal.
Depression Level | 1 year
  The Beck Depression Inventory (BDI) was used to determine the depression level of caregivers. The BDI was developed for measure the risk of depression, the level of depressive symptoms and changes in the severity of depression in adults. Reliability and validity of a Turkish version of the BDI were demonstrated by Hisli (1989). The BDI is a 21-item, self-rated scale and each item is scored between 1 and 3 points. Higher total scores indicate greater depression severity.
Anxiety Level | 1 year
  The Beck Anxiety Inventory (BAI) was used to evaluate the anxiety level of caregivers. The BAI was developed for determine the frequency of anxiety symptoms experienced by individuals. It is a 21-item, Likert scale with scores ranging from 0 and 3 points. Higher overall scores denote greater level of anxiety. Reliability and validity of a Turkish version of the BAI were demonstrated by Ulusoy et al. (1998).

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Yakut, Prof, Study Chair — Hasan Kalyoncu University
Locations (1):
- Serkan Usgu, Gaziantep, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is no plan for sharing

REFERENCES:
- [Result] Zhou J, Lin J, Leung WT, Wang L. A basic understanding of mucopolysaccharidosis: Incidence, clinical features, diagnosis, and management. Intractable Rare Dis Res. 2020 Feb;9(1):1-9. doi: 10.5582/irdr.2020.01011. PMID 32201668
- [Result] Guarany NR, Schwartz IV, Guarany FC, Giugliani R. Functional capacity evaluation of patients with mucopolysaccharidosis. J Pediatr Rehabil Med. 2012;5(1):37-46. doi: 10.3233/PRM-2012-0194. PMID 22543891
- [Result] Hendriksz CJ, Berger KI, Lampe C, Kircher SG, Orchard PJ, Southall R, Long S, Sande S, Gold JI. Health-related quality of life in mucopolysaccharidosis: looking beyond biomedical issues. Orphanet J Rare Dis. 2016 Aug 26;11(1):119. doi: 10.1186/s13023-016-0503-2. PMID 27561270
- [Result] Broomfield A, Davison J, Roberts J, Stewart C, Hensman P, Beesley C, Tylee K, Rust S, Schwahn B, Jameson E, Vijay S, Santra S, Sreekantam S, Ramaswami U, Chakrapani A, Raiman J, Cleary MA, Jones SA. Ten years of enzyme replacement therapy in paediatric onset mucopolysaccharidosis II in England. Mol Genet Metab. 2020 Feb;129(2):98-105. doi: 10.1016/j.ymgme.2019.07.016. Epub 2019 Jul 30. PMID 31383595
- [Result] Muenzer J. Early initiation of enzyme replacement therapy for the mucopolysaccharidoses. Mol Genet Metab. 2014 Feb;111(2):63-72. doi: 10.1016/j.ymgme.2013.11.015. Epub 2013 Dec 11. PMID 24388732